CLINICAL TRIAL: NCT03447574
Title: Non-invasive Fluid Volume During Fluid Shifts Technique Validation
Brief Title: Fluid Volume During Fluid Shifts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bruce Johnson, Consultant, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17-007104
Record Dates: First submitted 2018-02-16; First posted 2018-02-27 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Development of Non-invasive Protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim 1 (Experimental): The ethanol dilution is, in essence, a non-invasive dilution method. It is of interest because of how ethanol readily dissolves itself exclusively into the water space of the body[4], is non-toxic in reasonable concentrations, is metabolized in a 0th order reaction above concentrations of 0.015 g/dL[4], and there are non-invasive methods for determining blood alcohol concentration[5, 6]. Thus, by drinking a known amount of ethanol, total body water can be calculated after a few hours of periodic breathalyzer analyses. Ethanol has been validated against deuterium oxide, the invasive gold standard for determining total body water[4]. The ethanol dose will be 0.5g/kg body weight.
  Interventions: Other: ethanol dilution
- Aim 2 (Active Comparator): 30mL/kg body weight of saline will be rapidly infused after the baseline measurements completed in Aim 1. Non-invasive methods for fluid volume determination (CO-pulse-oximetry, ethanol breathalyzer, BIS) will be conducted and change from baseline calculated. To determine if non-invasive fluid volume techniques can accurately determine fluid changes in healthy participants.Non-invasive methods for fluid volume determination (CO-pulse-oximetry, ethanol breathalyzer, BIS) will be conducted and change from baseline calculated.
  Interventions: Other: ethanol dilution

INTERVENTIONS:
Other: ethanol dilution — Ethanol has been validated against deuterium oxide, the invasive gold standard for determining totally body water

SUMMARY:
This study is designed to answer the question of if several non-invasive methods are comparable to the invasive clinical gold standard of radiolabeled albumin in terms of detecting changes in fluid volume.

It is broken into two studies: Aim 1 Study A is designed as a pilot phase to develop the non-techniques, and Aim 2 Study B is comparing these techniques to the gold standard.

ELIGIBILITY:
1. Non-smokers
2. Have a BMI<30
3. Have no chronic disease
4. Be free of medications with known cardiovascular effects

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Validation against Gold Standard | 2 years
  The non-invasive methods being investigated will be non-inferior in measuring the blood or fluid volumes in healthy participants when compared to the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Johnson, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials